CLINICAL TRIAL: NCT06102941
Title: Cognitive Control Targets for the Treatment of Obsessive Compulsive Disorder in Young Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rachel Marsh, Principal Investigator, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAU8631; 1R61MH129544-01A1 (NIH)
Record Dates: First submitted 2023-10-16; First posted 2023-10-26 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Obsessive-Compulsive Disorder in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cognitive Training for Obsessive-Compulsive Disorder (Experimental): This is an open-label, one-arm study. Children who meet DSM-V diagnostic criteria for OCD and have clinically significant obsessive-compulsive symptoms (CY-BOCS score>16) will complete 4-weeks of at-home cognitive training.
  Interventions: Device: Cognitive Control Training (CT)

INTERVENTIONS:
Device: Cognitive Control Training (CT) — 4 weeks of an at-home computerized cognitive training program (AKL-T01) delivered on iPad (25 minutes/day, 5 days/week). Styled as a child-friendly video game, AKL-T01 CT taps focused attention, response inhibition, and working memory using a series of games with individually titrated difficulty to engage cognitive control processes.
  Other Names: AKL-T01; Akili

SUMMARY:
This study aims to examine the effects of a game-like program called cognitive control training (CT) for children with obsessive compulsive disorder (OCD). Children enrolled in this study will receive 4 weeks of the at-home computerized cognitive training program (AKL-T01) delivered on iPad (25 minutes/day, 5 days/week). Styled as a child-friendly video game, AKL-T01 CT taps focused attention, response inhibition, and working memory using a series of games to engage cognitive control processes. Children will complete the NIH Toolbox prior to, mid (2-weeks), and post-CT (4-weeks). Participants will complete MRI scans pre- and post-CT and then be offered a 12-week course of gold-standard Cognitive behavioral therapy with exposure and response prevention (or community referrals) after CT. The long-term goal of this study is to test how this CT intervention may enhance cognitive control capacity to reduce symptoms and improve response to cognitive behavioral therapy with exposure and response prevention in children with OCD.

DETAILED DESCRIPTION:
Obsessive-Compulsive Disorder (OCD) often onsets in childhood and, if not effectively treated, can lead to lifelong illness and poor functional outcomes. Cognitive behavioral therapy (CBT) with exposure and response prevention (EXRP) is the gold-standard, first-line treatment for children with OCD. However, as many as 40% of pediatric patients treated fail to remit. Based on the extant literature and our preliminary data showing that cognitive control functions are altered in children with OCD, this study is designed to test the hypothesis that cognitive control training (CT) should engage the Cognitive System to prime and augment EXRP response. A 2-year proof of concept study will be conducted to determine if CT enhances cognitive control behavioral performance (target engagement) in 60 children (8-12 years old) with OCD sampled from the general community and affiliated clinics. Children will receive 4 weeks of an at-home computerized cognitive training program (AKL-T01; FDA-approved for pediatric ADHD) delivered on iPad (25 minutes/day, 5 days/week). Styled as a child-friendly video game, AKL-T01 CT taps focused attention, response inhibition, and working memory using a series of games with individually titrated difficulty to engage cognitive control processes. Children will complete the NIH Toolbox prior to, mid (2-weeks), and post-CT (4-weeks). Cognitive control behavior will be indexed by NIH Toolbox Cognitive Function Composite. Participants will complete MRI scans pre- and post-CT and then be offered a 12-week course of gold-standard CBT EXRP (or community referrals) after CT. Resting state functional connectivity between task control networks and the Default Mode Network will be explored as a potential mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 8 and 12 years;
* Clinically significant OCD as the principal problem. This is defined as follows: they must meet DSM-V criteria for OCD as assessed with the Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children Present and Lifetime Version (K-SADS-PL). OCD must be the primary source of interference and distress (based on clinical evaluation with K- SADS-PL and Children's Yale-Brown Obsessive Compulsive Scale (C-YBOCS) and they must have clinically significant symptoms (i.e., C-YBOCS) ≥ 16;
* Not on psychotropic medication (either treatment-naïve or free of psychotropic medication for at least three months) and not receiving current psychotherapy for OCD;
* Ability to tolerate a treatment-free period (i.e., no treatment other than study CBT);
* Capacity to provide informed assent

Exclusion Criteria:

* Current or past diagnosis of major depressive disorder, PTSD, substance/alcohol abuse, psychotic disorder, bipolar disorder, eating disorder, pervasive developmental disorder, substance/alcohol dependence, or any other Axis I disorder not listed above;
* Active suicidal ideation;
* Females who are pregnant or nursing;
* Any major medical or neurological problem (e.g., unstable hypertension, seizure disorder, head trauma); -Positive urine screen for illicit drugs;
* Presence of metallic device or dental braces;
* IQ <80;

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
NIH Toolbox Cognition Battery | Baseline, 2-week follow-up (mid-training), and 4-week follow-up (post-training)
  Standardized Cognitive Function Composite Scores will be derived from the following NIH Toolbox tasks: 1) Flanker inhibitory control and attention task, 2) Dimensional Change Card Sort (DCCS) test of set-shifting function, 3) List of Working Memory Test, and 4) Pattern Comparison Processing Speed Test.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Marsh, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No